CLINICAL TRIAL: NCT00902213
Title: Physical Activity to Modify Sequelae and Quality of Life in Childhood Acute Lymphoblastic Leukemia: A Nursing Trial
Brief Title: Physical Activity to Modify Sequelae and Quality of Life in Childhood Acute Lymphoblastic Leukemia
Acronym: PAQOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PAQOL; R01CA129384 (NIH); NCI-2012-00017 (Registry Identifier: NCI Clinical Trial Registraiton Program)
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Physical Therapy Modalities; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minimal movement (No Intervention): Minimal movement group with usual care non-intervention.
- Physical Therapy (Active Comparator)
  Interventions: Behavioral: Physical Therapy; Behavioral: Support

INTERVENTIONS:
Behavioral: Physical Therapy — Each patient in this group will have physical therapy performed. The intervention will be tested for its effect on: 1) physical function outcomes (muscle strength, range of motion, endurance, gross motor skills), bone density and bone mineral content (end of therapy only); and 2) HRQL.
  Other Names: Physical Activity to Modify Sequelae and in Childhood ALL.
  Arms: Physical Therapy
Behavioral: Support — Visits with an Advanced Practice Nurse to support sustained motivation.
  Arms: Physical Therapy

SUMMARY:
This will be the first multidisciplinary, randomized, longitudinal trial of a tailored, parent- and child-focused physical activity program for children (ages 4- <19 years) with newly diagnosed ALL. It will test the ability of the intervention to prevent or diminish early physical function limitations and improve health-related quality of life (HRQL). The intervention will be tested for its effect on: 1) physical function outcomes (muscle strength, range of motion, endurance, gross motor skills), bone density and bone mineral content (end of therapy only); and 2) HRQL. This multi-site trial will test the intervention in 76 evaluable children with ALL (38 receiving the intervention and 38 receiving a placebo "minimal movement" standard care strategy).

DETAILED DESCRIPTION:
An advanced practice nurse (APN) will meet twice weekly with the patient and family for the first 4 weeks of the intervention to initiate the motivation-based dialogue and therapeutic interaction; this will be followed by once weekly visits during weeks 5-8 of the intervention; and monthly visits during weeks 9-through end of therapy. The physical therapist (PT) will meet at least once weekly with the patient and family during weeks 1-4 to initiate the prescriptive tailored exercise program; subsequent visits to reinforce and modify the program will occur at least once every other week during weeks 5-8, and at least once monthly during weeks 9-135 of the intervention. The PT will visit at least once weekly during weeks 1-4, at least once every other week during weeks 5-8, and at least once monthly during weeks 9-135. During weeks 9-135 of the intervention, the APN will call between the monthly in person-visits, if needed to those randomized to the MAP group to assure fidelity to the intervention and to provide booster support to the intervention where needed.

ELIGIBILITY:
Inclusion Criteria:

1. An immunophenotypic diagnosis of non-B cell ALL
2. Age 4 years through <19 years at diagnosis
3. 2-8 days on or per front line ALL treatment protocol
4. One parent or legal guardian (≥ 18 years) of the study subject who speaks and understands the English Language
5. Participant speaks and understands the English language
6. Written informed consent and child assent

Exclusion Criteria:

1. Age < 4 years or ≥19 years at diagnosis
2. A diagnosis of cerebral palsy or down syndrome
3. Second malignancy, chromosome breakage syndrome, or severe congenital immunodeficiency
4. Inability or unwillingness of research participant or legal guardian/representative to give written informed consent/assent
5. Females who are pregnant.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2009-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density/Bone Mineral Content | Assessed at baseline and at completion of therapy

SECONDARY OUTCOMES:
Health- related quality of life | Assessed at baseline, 8 and 15 weeks after baseline and at completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Cox, RN, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (4):
- United States (3):
  - AFLAC Cancer Center Children's Healthcare of Atlanta, Atlanta, Georgia
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - MD Anderson, Houston, Texas
- Toronto Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ness KK, Kaste SC, Zhu L, Pui CH, Jeha S, Nathan PC, Inaba H, Wasilewski-Masker K, Shah D, Wells RJ, Karlage RE, Robison LL, Cox CL. Skeletal, neuromuscular and fitness impairments among children with newly diagnosed acute lymphoblastic leukemia. Leuk Lymphoma. 2015 Apr;56(4):1004-11. doi: 10.3109/10428194.2014.944519. Epub 2014 Aug 20. PMID 25030039
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols